CLINICAL TRIAL: NCT00268112
Title: Resynchronization of Left Ventricular Contraction After Re-implantation of Anomalous Left Coronary Artery From the Pulmonary Artery (ALCAPA) Evaluated by Tissue Doppler Imaging
Brief Title: Resynchronization of Left Ventricular Contraction After Reimplantation of Anomalous Left Coronary Artery
Status: Terminated | Type: Observational
Why Stopped: sufficient data collected for analysis
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-203
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2006-12

CONDITIONS: Congenital Disorders
Keywords: pediatric; cardiac; ALCAPA; Tissue Doppler Imaging
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Bland White Garland Syndrome

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Spontaneous resynchronization of dyskinetic segments of the left ventricle occurs after coronary bypass surgery in adults and has been shown in some children. It is, however, unknown what degree of dyskinesis is likely to be reversible in infants with ischemia from anomalous coronary arteries and what criteria would indicate that a resynchronization strategy of biventricular pacing might be needed.

These questions need data from quantitative serial tissue Doppler observations of patients from pre-operative to late post-operative follow-up.

DETAILED DESCRIPTION:
We have previously studied, at Children's Healthcare of Atlanta, Egleston Hospital, 2 patients with ALCAPA and one other patient is currently enrolled in a prospective study after recent surgery, also at Children's Healthcare of Atlanta. We propose to study these 3 patients with this rare defect concurrently with their routine echocardiographic evaluations. Data will then be taken off-line for analysis.

Standard deviations of times to peak contraction velocity will be assessed for twelve cardiac segments. These will be reevaluated at follow up intervals after surgery on previously obtained echocardiograms. Those subjects in whom improvement of cardiac function, Left Ventricular Ejection Fraction (LVEF) and mitral regurgitation is seen will be compared to those in whom no improvement occurs.

ELIGIBILITY:
Inclusion Criteria:

* Re-implantation of an anomalous left coronary artery from the pulmonary artery

Exclusion Criteria:

* those patients who do not meet inclusion criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cardiac pediatric patients
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2004-01; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek A. Fyfe, MD, PhD, Principal Investigator — Sibley Heart Center Cardiology at Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States